CLINICAL TRIAL: NCT06626945
Title: AZAHAR Study. Observational Retrospective Study To Describe Characteristics And Clinical Outcomes of Patients With Systemic Lupus Erythematosus Initiating Saphnelo (Anifrolumab) in a Real-World Setting
Brief Title: AZAHAR Study To Describe Anifrolumab in a Real-World Setting
Acronym: AZAHAR
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3461R00080
Record Dates: First submitted 2024-09-26; First posted 2024-10-04 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
AZAHAR is an observational retrospective and longitudinal study with adults patients with SLE who initiated treatment with anifrolumab from June 1, 2023 to May 31, 2024.

The overall objective is to describe the characteristics and clinical outcomes of patients with SLE that initiated anifrolumab during its first year of commercialization in Spain.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic autoimmune disease characterized by altered immune response with excessive cytokines and antibodies production. Immune response activation and maintained inflammatory status promote a multisystemic dysfunction affecting numerous organs.

Anifrolumab, a monoclonal antibody that binds to type 1 IFN, which it is involved in pathways altered in SLE , blocks its effects. In clinical trials showed beneficial effects controlling the disease activity in patients with moderate and severe SLE, compared to standard of care. This biologic treatment was marketed in Spain on June 1, 2023. This study aims to describe real world evidence of anifrolumab in Spain since its commercialization.

The primary objective is to describe disease activity (including low disease activity state, (LLDAS)) and clinical remission at the initiation with anifrolumab and every 6 months, up to 18 months, after anifrolumab initiation.

The secondary objectives are:

1. To estimate the flare incidence rate, overall, and considering severe flares only, during the previous 12 months before anifrolumab initiation and every 6 months up to 18 months after anifrolumab initiation.
2. To describe SLE treatment, especially the use of corticosteroids (CS), during the previous 12 months before anifrolumab initiation, and every 6 months, up to 18 months after anifrolumab initiation.
3. To describe anifrolumab persistence and adherence rate over time during treatment with anifrolumab.
4. To describe healthcare resources utilization (HRU) for SLE during the previous 12 months before anifrolumab initiation and every 6 months, up to 18 months after anifrolumab initiation.

The exploratory objective is:

To describe organ damage at the anifrolumab initiation, and every 6 months, up to 18 months after anifrolumab initiation.

This is an observational retrospective and longitudinal chart review study including adults patients with moderate-severe SLE who initiated treatment with anifrolumab. Baseline data 12 months prior to anifrolumab treatment will be collected, and since anifrolumab initiation, participants will be followed-up until the closest available data to the end of the study (December 31st, 2024).

This study is based exclusively on secondary data collection from outpatient electronic medical records (EMRs). Therefore, it will rely on already existing data from patients by the time of data collection.

The expected sample size is around 120 patients from 20 hospitals in Spain.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilled the 2019 EULAR/ACR criteria for SLE at the date of anifrolumab initiation.
* Aged 18 years or older at the date of anifrolumab initiation.
* Have initiated anifrolumab between June 1st, 2023, and May 31st, 2024
* Have at least 12 months of medical history prior to anifrolumab initiation.

Exclusion Criteria:

* Current or previous exposure to anifrolumab as part of a clinical trial or Early Access Program (EAP).

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients diagnosed with SLE who attended the specialist's office at the participating hospitals in the study and initiated anifrolumab during the following period, between June 1st, 2023, and May 31st, 2024.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score | At anifrolumab initiation, and every 6 months after anifrolumab initiation, up to 18 months.
  The total score ranges between 0 and 105, with higher scores representing increased disease activity.
Physician Global Assessment (PGA) score | At anifrolumab initiation, and every 6 months after anifrolumab initiation, up to 18 months.
  PGA ranges from 0 to 3, with 0 representing the total inactivity of the disease and 3 an important activity.
  An increase of ≥1 score since the last visit is indicative of a flare.
Changes in SLEDAI-2K score | From anifrolumab initiation to 6, 12 and 18 months after anifrolumab initiation.
  Change from baseline in SLEDAI-2K score for consecutive timepoints.
Changes in PGA score | From anifrolumab initiation to 6, 12 and 18 months after anifrolumab initiation.
  Change from baseline in PGA score for consecutive timepoints.
Proportion of patients achieving low disease activity state | At anifrolumab initiation, and every 6 months after anifrolumab initiation, up to 18 months.
  LLDAS requires all the following criteria to be met:
  * SLEDAI-2K score ≤ 4, with no activity in the major organ systems (renal, central nervous system, cardiopulmonary, vasculitis, or fever).
  * No new SLEDAI-2K assessed disease activity compared to the previous visit.
  * PGA score ≤ 1
  * Prednisone or equivalent dosage ≤ 7.5 mg/day
  * No non-standard immunosuppressant dosing, with antimalarials allowed.
Proportion of patients achieving clinical remission | At anifrolumab initiation, and every 6 months after anifrolumab initiation, up to 18 months.
  Clinical remission will be measured as DORIS-21, a composite endpoint including:
  * Clinical SLEDAI score of 0 (no disease activity)
  * PGA <0.5
  * Prednisolone dose of 5 mg/day or less.
  * Stable use of antimalarials, immunosuppressives, and biologics.

SECONDARY OUTCOMES:
Flares incidence rate | 12 months before anifrolumab initiation and every 6 months after anifrolumab initiation, up to 18 months.
  Flares is defined as worsening of symptoms based as assessed with a modified revised Safety of Estrogens in Lupus National Assessment-Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI) flare index (rSFI) based on SLEDAI-2K assessment.
Anifrolumab adherence | Up to 18 months since anifrolumab initiation.
  Proportion of anifrolumab infusions that happen every 18 to 38 days during a certain specified period from first anifrolumab infusion.
Anifrolumab persistence | Up to 18 months since anifrolumab initiation.
  Time on treatment until discontinuation or end of follow-up
Proportion of patients receiving any of dose of corticosteroids (CS) | Previous 12 months before anifrolumab initiation, and every 6 months after anifrolumab initiation, up to 18 months.
  CS include the following route of administration: oral, subcutaneous, intramuscular or intravenous.
Annual cumulative dose of CS | Previous 12 months before anifrolumab initiation, and every 6 months after anifrolumab initiation, up to 18 months
  Corticosteroids include the following route of administration: oral, subcutaneous, intramuscular or intravenous.
Proportion of patients treated with any biologic treatment | Previous 12 months before anifrolumab initiation.
  Biologic treatment refers to any biologic medication (on-label and off-label) prescribed for SLE.
Proportion of patients treated with any antimalarial medication | Previous 12 months before anifrolumab initiation and every 6 months after anifrolumab initiation, up to 18 months after anifrolumab initiation.
  Antimalarial medication prescribed for SLE.
Proportion of patients treated with any immunosuppressive medication | Previous 12 months before anifrolumab initiation and every 6 months after anifrolumab initiation, up to 18 months after anifrolumab initiation.
  Immunosuppressive medication prescribed for SLE.
Hospitalization rate attributable to SLE | Previous 12 months before anifrolumab initiation and every 6 months after anifrolumab initiation, up to 18 months after anifrolumab initiation.
  Annual hospitalization rate expressed by patient-year
Intensive care unit (ICU) admission rate attributable to SLE | Previous 12 months before anifrolumab initiation and every 6 months after anifrolumab initiation, up to 18 months after anifrolumab initiation.
  Annual ICU admission rate expressed by patient-year
Emergency room (ER) admission rate attributable to SLE | Previous 12 months before anifrolumab initiation and every 6 months after anifrolumab initiation, up to 18 months after anifrolumab initiation.
  Annual ED admission rate expressed by patient-year
Primary care (PC) visits rate attributable to SLE | Previous 12 months before anifrolumab initiation and every 6 months after anifrolumab initiation, up to 18 months after anifrolumab initiation.
  Annual PC visits rate expressed by patient-year
Specialist visits rate attributable to SLE | Previous 12 months before anifrolumab initiation and every 6 months after anifrolumab initiation, up to 18 months after anifrolumab initiation.
  Annual specialist visits rate expressed by patient-year

OTHER OUTCOMES:
SLICC/ACR (Systemic Lupus International Collaborating Clinics/American College of Rheumatology) Damage Index for SLE (SDI) score | At anifrolumab initiation and every 6 months after anifrolumab initiation, up to 18 months.
  SDI contains items that should be present for at least 6 months with the exception that manifestations such as myocardial infarction and stroke are recorded once they occur. Damage is defined for 12 organ systems: ocular (range 0-2), neuropsychiatric (0-6), renal (0-3), pulmonary (0-5), cardiovascular (0-6), peripheral vascular (0-5), gastrointestinal (0-6), musculoskeletal (0-7), skin (0-3), endocrine (diabetes) (0-1), gonadal (0-1), and malignancies (0-2). Damage over time can only be stable or increase, theoretically to a maximum of 47 points. Higher scores indicate higher organ damage.
Change in SDI score | From anifrolumab initiation to 6, 12 and 18 months after anifrolumab initiation.
  Change from baseline in SDI score for consecutive timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Josefina Cortés-Hernández, MD, PhD, Principal Investigator — Unit of Lupus, VHIR-Hospital Universitary Vall d'Hebrón
Locations (13):
- Spain (13):
  - Research Site, Barcelona
  - Research Site, Granada
  - Research Site, Jaén
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, León
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Mérida
  - Research Site, Móstoles
  - Research Site, Murcia
  - Research Site, Seville
  - Research Site, Toledo
  - Research Site, Valladolid

REFERENCES:
- [Derived] Galindo-Izquierdo M, Bahamontes-Rosa N, Sarto-Ferres B, Galvez-Fernandez M, Cortes-Hernandez J. Characteristics and clinical outcomes of patients with systemic lupus erythematosus initiating anifrolumab in a real-world setting in Spain (AZAHAR study): an observational study protocol. Lupus Sci Med. 2025 Feb 12;12(1):e001486. doi: 10.1136/lupus-2024-001486. PMID 39939126